CLINICAL TRIAL: NCT07384637
Title: Effects of Progressive Relaxation Exercises and Planned Training After Cesarean Section on Pain, Anxiety and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Sukran Ertekin Pinar, Prof. Dr., Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR SİVAS 07; SFF-2022-096 (Other Grant/Funding Number: Sivas Cumhuriyet University Scientific Research Projects)
Record Dates: First submitted 2026-01-27; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2023-01

CONDITIONS: Relaxation Exercises and Training After Cesarean Section
Keywords: Caesarean, Pain, Anxiety, Comfort, Exercise, Education
MeSH Terms: conditions — Pain; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Progressive Relaxation Exercises after Cesarean Section (Experimental): Progressive relaxation exercises began with breathing exercises, continued with muscle relaxation exercises, and lasted 30 minutes. Before starting the exercise, the environment was made quiet and free from external disturbances. The patient was also seated comfortably, and standard meditation music was played during the exercise. Progressive relaxation exercises combine the contraction and relaxation of large muscle groups such as the face, arms, legs, neck, and back with deep breathing. The exercises were performed by taking a deep breath, tensing the muscles, maintaining this tension for 5-7 seconds, and then relaxing the muscles (15-20 seconds). Throughout the exercise, the individual was instructed to continue breathing slowly and deeply through the nose and exhaling through the mouth.
  Interventions: Behavioral: Progressive Relaxation Exercise group
- Planned Training after Cesarean Section (Experimental): The training group received pre-planned training based on the literature. The training content included topics such as postpartum uterine changes, bleeding and vaginal discharge, elimination, sleep and rest, postpartum blues, medication use, initiation of sexual intercourse, timing of the resumption of menstruation, contraceptive methods, nutrition, breast care and breast problems, infant care, breastfeeding, and infant vaccinations. During the training, educational materials such as illustrated guides on family planning were used, and an educational brochure prepared by the researcher based on the literature was also given to the women after the training. The training was conducted face-to-face with each woman by the researcher, in accordance with adult education principles, and lasted 30-45 minutes. In addition, training methods such as lecturing, question-and-answer, discussion, brainstorming, and problem-solving were used during the training.
  Interventions: Behavioral: Planned Education group
- Standard of care Group (No Intervention): The control group received no treatment. They only received standard hospital care procedures along with the Visual Analog Scale, State-Trait Anxiety Inventory, and Postpartum Comfort Scale (pre-test, post-test).

INTERVENTIONS:
Behavioral: Progressive Relaxation Exercise group — On the first postoperative day, the women were met with, informed, and their written consent was obtained. Women in the Progressive Relaxation Exercise group who met the inclusion criteria were administered the Personal Information Form, Visual Analog Scale, State-Trait Anxiety Inventory, and Postpartum Comfort Scale via face-to-face interviews on the first postoperative day. Completing all forms took 15-20 minutes. Relaxation exercises began with breathing exercises, continued with muscle relaxation exercises, and lasted 30 minutes. In the final test phase, the Visual Analog Scale, State-Trait Anxiety Inventory, and Postpartum Comfort Scale were repeated on the second postoperative day.
  Arms: Progressive Relaxation Exercises after Cesarean Section
Behavioral: Planned Education group — On the first postoperative day, the women were met with, informed, and their written consent was obtained. Women in the Planned Education group who met the inclusion criteria were administered the Personal Information Form, Visual Analog Scale, State-Trait Anxiety Inventory, and Postpartum Comfort Scale via face-to-face interviews on the first day. Completing all forms took 15-20 minutes. The training was conducted face-to-face by the researcher for each woman, in accordance with adult education principles, and lasted 30-45 minutes.
  Arms: Planned Training after Cesarean Section

SUMMARY:
Effects of Progressive Relaxation Exercises and Planned Training after Cesarean Section on Pain, Anxiety and Comfort

DETAILED DESCRIPTION:
The study consisted of a total of 129 women who underwent cesarean section (progressive relaxation exercise group: 43, planned training group: 43, control group: 43). Data were collected using a Personal Information Form, Visual Analog Scale, State-Trait Anxiety Inventory, and Postpartum Comfort Scale. Intergroup comparisons revealed statistically significant differences (p˂0.05) in the mean scores of the Visual Analog Scale, State Anxiety Inventory, Trait Anxiety Inventory, and Postpartum Comfort Scale in the post-test after exercise and training for women in the exercise, training, and control groups. After progressive relaxation exercise and training, pain levels decreased in women in the exercise and training groups, anxiety levels decreased in women in the training group, and comfort levels increased in women in both the exercise and training groups.

ELIGIBILITY:
Inclusion Criteria:

* on the first postoperative day,
* at least four hours after analgesic administration,
* mobilized,
* with their baby present,
* their baby without any health problems,
* without any physical or mental illness,
* without communication problems,
* who volunteered to participate were included in the study.

Exclusion Criteria:

* women who were not present on the first postoperative day,
* had not received analgesic treatment for at least four hours,
* were not mobile,
* did not have their baby with them,
* their baby had any health problems,
* they had a physical or mental illness,
* they had difficulty communicating,
* they did not volunteer to participate were excluded from the study.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | baseline
  The scale is graded as 0-10 cm long, with 0=no pain, 10=the most severe pain. It is applied by the individual marking a point corresponding to the level of pain they feel. The distance between the determined point and the lowest part of the line is evaluated in centimeters. The value found indicates the patient's pain level.
State-Trait Anxiety Inventory | Baseline
  The State Anxiety Inventory consists of 20 items and requires individuals to describe how they feel at a specific moment under specific circumstances, taking into account their feelings about the situation. The Trait Anxiety Inventory also consists of 20 items and requires individuals to describe how they feel in a given situation, regardless of the circumstances. High scores on both the State and Trait Anxiety Inventories indicate high anxiety levels, while low scores indicate low anxiety levels.
Postpartum Comfort Scale | Baseline
  The Postpartum Comfort Scale assesses the physical, psychospiritual, and sociocultural comfort of women who have had both cesarean and vaginal deliveries. Physical and bodily perceptions constitute the physical comfort subscale. Spiritual and psychological components form the psychospiritual comfort subscale. Interpersonal, family, and social relationships, as well as components related to finances and support systems, constitute the sociocultural comfort subscale. The scale, which uses a five-point Likert scale, consists of 34 items. The lowest possible score is 34, and the highest is 170. Values close to 170 indicate a high level of comfort.

SECONDARY OUTCOMES:
Visual Analog Scale | On the second postoperative day after a cesarean section
  The scale is graded as 0-10 cm long, with 0=no pain, 10=the most severe pain. It is applied by the individual marking a point corresponding to the level of pain they feel. The distance between the determined point and the lowest part of the line is evaluated in centimeters. The value found indicates the patient's pain level.
State-Trait Anxiety Inventory | On the second postoperative day after a cesarean section
  The State Anxiety Inventory consists of 20 items and requires individuals to describe how they feel at a specific moment under specific circumstances, taking into account their feelings about the situation. The Trait Anxiety Inventory also consists of 20 items and requires individuals to describe how they feel in a given situation, regardless of the circumstances. High scores on both the State and Trait Anxiety Inventories indicate high anxiety levels, while low scores indicate low anxiety levels.
Postpartum Comfort Scale | On the second postoperative day after a cesarean section
  The Postpartum Comfort Scale assesses the physical, psychospiritual, and sociocultural comfort of women who have had both cesarean and vaginal deliveries. Physical and bodily perceptions constitute the physical comfort subscale. Spiritual and psychological components form the psychospiritual comfort subscale. Interpersonal, family, and social relationships, as well as components related to finances and support systems, constitute the sociocultural comfort subscale. The scale, which uses a five-point Likert scale, consists of 34 items. The lowest possible score is 34, and the highest is 170. Values close to 170 indicate a high level of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Sukran Ertekin Pinar, Prof. Dr., Principal Investigator — Cumhuriyet University
Locations (1):
- Sivas Cumhuriyet University, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No